CLINICAL TRIAL: NCT04178330
Title: Tomotherapy as Primary Radiotherapy for Multipule Brain Metastases:A Single Arm, Single Center,Phase II Trial
Brief Title: Tomotherapy as Primary Radiotherapy for Multipule Brain Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianping Xiao, Dr, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2014 YZ-14-01
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Brain Metastases
Keywords: multiple brain metastases; Tomotherapy; fractionated stereotactic radiotheray
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): patients with multiple brain metastases (no less than 3 lesions) ,who have not recived whole brain radiotheray (WBRT).
  Interventions: Radiation: tomotherapy

INTERVENTIONS:
Radiation: tomotherapy — Whole brain radiation (WBRT) with 38-40Gy in 20 fractions and concurrent boost of 60-70Gy of the lesions. TMZ is used if necessary: concomitant TMZ: 75mg/m2 adjuvant TMZ: 150mg/ m2*5d, q28d, up to 6cycles.

SUMMARY:
This clinical trial was designed to investigate the efficiency and toxicity of tomotherapy as primary radiotherapy for multiple brain metastases.

DETAILED DESCRIPTION:
This is a single-arm, single center, phase II trial to investigate the feasibility and toxicity of tomotherapy as primary radiotherapy for multiple brain metastases(≥3 lesions).

ELIGIBILITY:
Inclusion Criteria:Histologic or cytologic diagnosis of primary tumor and conformed brain metastases by enhanced MRI or CT; the lesion number is no less than 3;KPS ≥60,or KPS ≥40 and the limitation of motion is simply caused by brain tumor that is adjacent to the motor function areas; Age: 18-75 years old; Adequate organ function:WBC≥4.0x109/L, Neu ≥ 1.5x109/L, Hemoglobin ≥ 110 g/L, Platelets ≥100 x109/L, Totalbilirubin ≤ 1.5x ULN, AST and ALT ≤ 1.5x ULN, BUN and Cr: within the normal range.

Exclusion Criteria: Other clinically significant diseases (e.g.myocardial infarction within the past 6 months, severe arrhythmia). Unable or unwilling to comply with the study protocol.The expected survival time is less than 3 months. Patients who are anticipated in other clinical trials of brain metastases. Patients who has been treated with WBRT. Pregnant patients or female patients whose HCG is positive. Unsuitable to participate in study, that in the opinion of the treating physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Disease control rate(DCR) | 2-3 month after radiation
  Using RTOG9508 criteria, tumor control is defined as CR+PR+SD

SECONDARY OUTCOMES:
Overall survival | up to 3 years
  the time from radiation to death
progress free survival | up to 1 year
  the time from radiation to any progression
local control rate | up to 1 year
  the time from radiation to the treated brain metastases recurrence
intracranial progress free survival rate | up to 1 year
  the time from radiation to local recurrence and/or new brain metastases
adverse event | from the day of radiation, up to 3 years
  acute and late toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Xiao, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No